CLINICAL TRIAL: NCT01704456
Title: Integrated Mindfulness-based Cognitive Behaviour Therapy Versus Cognitive Behaviour Therapy for Provoked Vestibulodynia
Acronym: COMFORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Lori Brotto, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H12-02358
Record Dates: First submitted 2012-08-22; First posted 2012-10-11 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-02

CONDITIONS: Provoked Vestibulodynia
Keywords: provoked vestibulodynia; dyspareunia; vulvodynia; mindfulness; cognitive behavioural therapy
MeSH Terms: conditions — Dyspareunia; Vulvodynia | interventions — Mindfulness-Based Cognitive Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-based cognitive therapy (MBCT) (Experimental): Women in the MBCT Group Treatment arm will receive the treatment in small group format (8-9 women). Each session will be 2.25 hours in duration and there will be eight, weekly sessions over the course of 2 months. Session content includes education about chronic pain, PVD, stress and sexual response, mindfulness practices, and cognitive techniques to notice thought patterns that contribute to increased pain.
  Interventions: Behavioral: Mindfulness-based Cognitive Therapy
- Cognitive Behavioural Therapy (CBT) (Experimental): Women in the CBT Group Treatment arm will receive the treatment in small group format (8-9 women). Each session will be 2.25 hrs in duration and there will be eight, weekly sessions over the course of 2 months. Session content includes education about chronic pain, PVD, stress and sexual response, behavioural techniques such as progressive muscle relaxation, cognitive techniques to challenge unhealthy thinking patterns, and communication skills training.
  Interventions: Behavioral: Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Mindfulness-based Cognitive Therapy — The MBCT intervention will be administered in small group format (8-9 women). Each session will be 2.25 hours in duration and there will be eight, weekly sessions over the course of 2 months. Session content includes education about chronic pain, PVD, stress and sexual response, mindfulness practices, and cognitive techniques to notice thought patterns that contribute to increased pain.
  Other Names: MBCT
  Arms: Mindfulness-based cognitive therapy (MBCT)
Behavioral: Cognitive Behavioural Therapy — The CBT intervention will be administered to women in small group format (8-9 women). Each session will be 2.25-hrs in duration and there will be eight, weekly sessions over the course of 2 months. Session content includes education about chronic pain, PVD, stress and sexual response, behavioural techniques such as progressive muscle relaxation, cognitive techniques to challenge unhealthy thinking patterns, and communication skills training.
  Other Names: CBT
  Arms: Cognitive Behavioural Therapy (CBT)

SUMMARY:
This randomized trial, nicknamed the COMFORT (Cognitive therapy or Mindfulness FOR Treatment of pvd) study, will compare the effects of an 8-session group Mindfulness-based Cognitive Therapy (MBCT) to an 8-session group Cognitive Behavioural Therapy (CBT) for women with provoked vestibulodynia (PVD). Women with PVD will be randomly assigned to attend either eight sessions of group MBCT or CBT. Each session is 2.25 hours long and spaced 1 week apart. The purpose of this study is to determine whether the 8-session MBCT intervention for PVD is no worse than an 8-session CBT intervention for decreasing women's pain intensity, sexual distress, catastrophizing and hypervigilance towards pain.

DETAILED DESCRIPTION:
PURPOSE:

The purpose of this study is to determine whether an 8-session MBCT intervention for PVD is no worse than an 8-session CBT intervention for improving women's pain intensity and reducing their sexual distress, catastrophizing and hypervigilance towards pain. The investigators will also examine whether pain improvements at follow-up are mediated by changes in self-compassion and mindfulness (in the MBCT arm only) and moderated by pre-treatment credibility, personality, and anxiety sensitivity.

HYPOTHESES:

1. At follow-up (4 weeks, 6 months and 12 months post-treatment), women in the MBCT arm will experience a greater decline (vs. pre-treatment) in vestibular pain intensity compared to women in the CBT arm.
2. At follow-up (4 weeks, 6 months and 12 months post-treatment), women in the MBCT arm will experience a greater decline (vs. pre-treatment) in sex-related distress, pain catastrophizing, hypervigilance, and self-reported pain during intercourse/other penetrative sex compared to women in the CBT arm.
3. The investigators hypothesize that improvements in pain intensity during vestibular touch will be mediated by changes in self-compassion and mindfulness in the MBCT arm only at 6 and 12 months follow-up.
4. The investigators hypothesize that pre-treatment credibility, personality, and anxiety sensitivity will significantly moderate improvements in pain intensity during vestibular touch at 6 and 12 months follow-up.
5. The investigators hypothesize improvements in both arms on the "Patient Global Impression of Change Scale" and significantly greater improvements in the MBCT arm relative to the CBT arm at follow-up (4 weeks, 6 months and 12 months post-treatment).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of provoked vestibulodynia (PVD)
* 19 years of age or older
* premenopausal
* fluent in English
* during the study, women must agree not to change any medications they are taking for PVD.

Exclusion Criteria:

* unprovoked vulvar pain, other pathology causing pain with penetration, or chronic pelvic pain
* being uncomfortable and unwilling to participate in a group setting.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-10; Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Brotto, PhD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - British Columbia Centre for Sexual Medicine, Vancouver, British Columbia
  - Department of Gynaecology, Vancouver, British Columbia

REFERENCES:
- [Derived] Brotto LA, Zdaniuk B, Rietchel L, Basson R, Bergeron S. Moderators of Improvement From Mindfulness-Based vs Traditional Cognitive Behavioral Therapy for the Treatment of Provoked Vestibulodynia. J Sex Med. 2020 Nov;17(11):2247-2259. doi: 10.1016/j.jsxm.2020.07.080. Epub 2020 Aug 22. PMID 32843320
- See also: UBC Sexual Health Lab — http://brottolab.med.ubc.ca
- See also: Published Paper — https://med-fom-brotto.sites.olt.ubc.ca/files/2019/07/Brotto-et-al.-A-comparison-of-mindfulness2019.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness-based Cognitive Therapy (MBCT) | Cognitive Behavioural Therapy (CBT)
Started | 67 | 63
Completed | 59 | 49
Not Completed | 8 | 14
Not completed — Lost to Follow-up | 8 | 14

BASELINE CHARACTERISTICS:
Population: Participants comprised a total of 130 women diagnosed with PVD by a physician.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness-based Cognitive Therapy (MBCT) | Cognitive Behavioural Therapy (CBT) | Total
Number analyzed (Participants) | 67 | 63 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.72 (7.48) | 31.24 (8.99) | 32.35 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 63 | 130
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Euro-Canadian | 46 | 38 | 84
  South/East Asian | 10 | 11 | 21
  Other | 9 | 12 | 21
  Prefer Not To Answer | 2 | 2 | 4
Relationship status [Count of Participants; unit: Participants]
  Married / Common Law | 45 | 41 | 86
  Dating | 11 | 13 | 24
  Single | 11 | 8 | 19
  Did Not Disclose | 0 | 1 | 1
Length of relationship [Mean (Standard Deviation); unit: years] | 7.77 (6.16) | 7.56 (6.79) | 7.67 (7.52)
Satisfaction with relationship closeness (/10) [Mean (Standard Deviation); unit: units on a scale] — How satisfied are you with the level of closeness in your relationship on a scale where 0=completely dissatisfied and 10=completely satisfied
  units on a scale | 7.26 (2.29) | 7.79 (1.99) | 7.52 (2.15)
Education [Number; unit: participants]
  High School | 1 | 2 | 3
  Some College | 10 | 17 | 27
  University Degree | 31 | 24 | 55
  Post-Graduate | 17 | 13 | 30
  Prefer Not To Answer | 8 | 7 | 15
Level of typical pain (/10) [Mean (Standard Deviation); unit: units on a scale] — Numeric Rating Scale that asked participants to rate the "intensity of pain during vaginal penetration attempts with sexual intercourse or penetration over the past 4 weeks." This question was rated on a 0 to 10 scale from no pain (0) to worst possible pain (10).
  units on a scale | 6.04 (1.82) | 5.96 (2.11) | 6.00 (1.96)
Level of worst pain (/10) [Mean (Standard Deviation); unit: units on a scale] — Numeric Rating Scale that asked participants to rate the "intensity of pain during vaginal penetration attempts with sexual intercourse or penetration over the past 4 weeks" This question was rated on a 0 to 10 scale from no pain (0) to worst possible pain (10)
  units on a scale | 8.23 (1.10) | 8.23 (1.32) | 8.23 (1.21)
Years since diagnosis [Mean (Standard Deviation); unit: years] | 9.85 (7.72) | 6.02 (4.72) | 7.95 (6.67)
PVD history [Count of Participants; unit: Participants] — Lifelong vs Aquired PVD
  Participants
    Lifelong | 43 | 37 | 80
    Aquired | 24 | 26 | 50
Past treatments received [Number; unit: participants] | 36 | 29 | 65
Past medications received [Number; unit: participants] | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Vulvslgesiometer Pain Rating From Baseline to One Month Post-treatment to 6 Months Post-treatment
Description: The investigators have selected pain intensity during a controlled examination as the primary endpoint in this study. Specifically, pain intensity at the vulvar vestibule will be assessed using a vulvalgesiometer. The vulvalgesiometer is an instrument that provides a measure of pain/sensitivity that can be standardized across time points. The vulvalgesiometer is calibrated to exert a fixed amount of pressure. In this study, 30 grams of pressure at the 1, 3, 4, 6, 8, 9, and 11 o'clock positions (randomly) around the vestibule will be applied using the vulvalgestiometer. Women will also report their pain at each site using a numeric rating scale from 0 (no pain) to 10 (worst pain ever).
Time Frame: Pre-treatment, one month post-treatment and 6 months post-treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Cognitive Therapy (MBCT) | Cognitive Behavioural Therapy (CBT)
Number analyzed (Participants) | 67 | 63
score on a scale
  pre-treatment | 6.66 (2.17) | 6.62 (2.19)
  one month post-treatment | 3.21 (1.96) | 3.60 (2.14)
  6 months follow up | 2.92 (2.31) | 2.86 (1.89)

2. Secondary Outcome: Self-reported Pain During Penetration
Description: The investigators will measure self-report of pain during attempted or completed intercourse (or dildo entry for non-heterosexual women). Numeric Rating Scale that asked participants to rate the "intensity of pain during vaginal penetration attempts with sexual intercourse or penetration over the past 4 weeks" This question was rated on a 0 to 10 scale from no pain (0) to worst possible pain (10).
Time Frame: Pre-treatment,one month post-treatment, and 6 months follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Cognitive Therapy (MBCT) | Cognitive Behavioural Therapy (CBT)
Number analyzed (Participants) | 67 | 63
score on a scale
  Pre-treatment | 6.69 (1.91) | 5.86 (2.13)
  One Month Post-Treatment | 4.34 (2.22) | 4.65 (2.21)
  6 months follow up | 3.39 (1.89) | 4.03 (2.11)

3. Secondary Outcome: Sexual Function
Description: The investigators will examine women's self-reported sexual function by administering the Female Sexual Function Index (FSFI). The Female Sexual Function Index (FSFI) is a 19-item self-report questionnaire which assesses sexual function in women. It covers six sexual domains: lubrication, arousal, desire, pain, orgasm and satisfaction. Scores range from 7.2 - 36 where increase in sexual dysfunction is represented by lower scores.
  Subscales:
  Desire- 2, 3 [Subscale scores Range: 1.2 - 6] Arousal- 5,6,7,8 [Subscale Scores Range: 1.2 - 6] Lubrication- 9,10,11,12 [Subscale Scores Range: 1.2 - 6] Orgasm- 13, 14, 15 [Subscale Scores Range: 1.2 - 6] Satisfaction- 1, 16, 17 [Subscale Scores Range: 1.2 - 6] Pain- 18, 19, 20 [Subscale Scores Range: 1.2 - 6] Extra item: (4) have you been sexually active in past 4 weeks? (yes/no) [Scores Range 0 (no) - 1 (yes)]
  Note: Ranges applicable only if question 4 was answered "yes".
Time Frame: Pre-treatment, one month post-treatment, and 6 months post-treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Cognitive Therapy (MBCT) | Cognitive Behavioural Therapy (CBT)
Number analyzed (Participants) | 67 | 63
score on a scale
  Pre-Treatment | 19.57 (6.29) | 21.18 (6.10)
  One Month Post-Treatment | 21.79 (6.83) | 23.41 (5.72)
  6 months follow up | 24.75 (5.62) | 23.20 (5.45)

4. Secondary Outcome: Sexual Distress
Description: The investigators will examine women's self-reported sexual distress by administering the Female Sexual Distress Scale-Revised. This is a 12-item self-report questionnaire assessing for sexuality related personal distress. Scores on the scale range from 0 - 48, where higher scores represent higher levels of distress.
Time Frame: Pre-treatment, one month post-treatment, and 6 months post-treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Cognitive Therapy (MBCT) | Cognitive Behavioural Therapy (CBT)
Number analyzed (Participants) | 67 | 63
score on a scale
  Pre-Treatment | 34.28 (11.18) | 35.68 (10.43)
  One Month Post-Treatment | 26.60 (13.35) | 24.93 (91.31)
  6 months follow up | 22.81 (12.98) | 23.77 (9.61)

5. Secondary Outcome: Pain Catastrophizing
Description: The investigators will examine women's self-reported pain catastrophizing by administering the Pain Catastrophizing Scale. The Pain Catastrophizing Scale (PCS) is a self-report questionnaire that asks participants to think about past painful experiences, or a specific experience of pain, and to indicate the degree to which they have any of the presented thoughts or feelings when they are experiencing pain. Each one of the 13-items is rated on a Likert scale from 0 (not at all) to 4 (all the time), where a higher total score indicates higher pain catastrophizing.
  Subscales: Rumination- (4 items) 8, 9, 10, and 11 [Scores Range: 0 - 16] Magnification- (3 items) 6, 7, and 13 [Scores Range: 0 - 12] Helplessness- (6 items) 1, 2, 3, 4, 5, and 12 [Scores Range: 0 - 24] Sum of all items [Overall Range: 0 - 52]
Time Frame: Pre-treatment, one month post-treatment, and 6 months post-treatment..
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Cognitive Therapy (MBCT) | Cognitive Behavioural Therapy (CBT)
Number analyzed (Participants) | 67 | 63
score on a scale
  Pre-Treatment | 26.92 (12.86) | 25.62 (11.97)
  One Month Post-Treatment | 15.64 (12.54) | 12.57 (8.13)
  6 months follow up | 11.55 (9.91) | 10.83 (7.66)

6. Secondary Outcome: Pain Hypervigilance
Description: The investigators will examine women's self-reported hypervigilance about pain by administering the Pain Vigilance and Awareness Questionnaire. The Pain Vigilance and Awareness Questionnaire (PVAQ) is a 16 item self-report measure to assess the awareness, vigilance, preoccupation and observation of pain. Sum total score [Scores Range: 0 - 80].
Time Frame: Pre-treatment, one month post-treatment, and 6 months post treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Cognitive Therapy (MBCT) | Cognitive Behavioural Therapy (CBT)
Number analyzed (Participants) | 67 | 63
score on a scale
  Pre-Treatment | 43.24 (14.67) | 42.46 (12.12)
  One Month Post-Treatment | 39.74 (13.72) | 40.32 (14.19)
  6 months follow up | 38.50 (13.88) | 38.76 (14.47)

7. Secondary Outcome: Chronic Pain Acceptance, Activities Engagement
Description: The investigators will examine women's self-reported pain acceptance, activities engagement, by administering the CPAQ chronic pain acceptance questionnaire. The Chronic Pain Acceptance Questionnaire (CPAQ) measures the degree of acceptance of pain by chronic pain patients. It consists of 20 items measuring two domains, Activities Engagement and Pain Willingness. Total score range is from 0 - 120, with higher scores indicating higher levels of pain acceptance.
  Subscales:
  Activities engagement (11 items)- Q 1, 2, 3, 5, 6, 8, 9, 10, 12, 15, 19 [Scores Range: 0 - 66] Pain willingness (9 items)- Q 4, 7, 11, 13, 14, 16, 17, 18, 20 [Scores Range: 0 - 54]
Time Frame: Pre-treatment, one month post-treatment, and 6 months post-treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Cognitive Therapy (MBCT) | Cognitive Behavioural Therapy (CBT)
Number analyzed (Participants) | 67 | 63
score on a scale
  Pre-Treatment | 42.40 (10.91) | 42.39 (10.14)
  One Month Post-Treatment | 47.97 (10.26) | 46.63 (9.34)
  6 months follow up | 49.24 (9.29) | 47.83 (8.70)

8. Secondary Outcome: Chronic Pain Acceptance, CPAQ Pain Willingness
Description: The investigators will examine women's self-reported pain acceptance, activities engagement, by administering the CPAQ chronic pain acceptance questionnaire. The Chronic Pain Acceptance Questionnaire (CPAQ) measures the degree of acceptance of pain by chronic pain patients. It consists of 20 items measuring two domains: Activities Engagement and Pain Willingness. Total score range is from 0 - 120, with higher scores indicating higher levels of pain acceptance.
  Subscales:
  Activities engagement (11 items)- Q 1, 2, 3, 5, 6, 8, 9, 10, 12, 15, 19 [Scores Range: 0 - 66] Pain willingness (9 items)- Q 4, 7, 11, 13, 14, 16, 17, 18, 20 [Scores Range: 0 - 54]
Time Frame: Pre-treatment, one month post-treatment, and 6 months post treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Cognitive Therapy (MBCT) | Cognitive Behavioural Therapy (CBT)
Number analyzed (Participants) | 67 | 63
score on a scale
  Pre-Treatment | 23.99 (9.29) | 22.91 (8.05)
  One Month Post-Treatment | 29.34 (10.07) | 29.20 (8.42)
  6 months follow up | 33.72 (8.80) | 31.29 (8.51)

ADVERSE EVENTS:
Time Frame: The entire duration of the study up to 6 months post treatment.
Description: Adverse event data was not collected; only reason for withdrawal. We interpreted risk as being due to a medication and this was a behavioral trial. We did not exclude participants with symptoms of anxiety or depression, and it is possible that those symptoms may have put participants at risk.
Arm/Group | Mindfulness-based Cognitive Therapy (MBCT) | Cognitive Behavioural Therapy (CBT)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No